CLINICAL TRIAL: NCT01140594
Title: A Prospective Randomized Eye to Eye Comparison of Fellow Eyes Undergoing Lasik With the IntraLase(TM) FS Versus PRK
Brief Title: Wavefront-guided Photorefractive Keratectomy (PRK) Versus Wavefront-guided Lasik for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SU-05192010-6082; SQL 97234
Record Dates: First submitted 2010-06-02; First posted 2010-06-09 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Photorefractive Keratectomy; Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront-guided PRK (Active Comparator): Wavefront-guided PRK
  Interventions: Procedure: Photorefractive keratectomy; Procedure: Laser in-situ keratomileusis
- Wavefront-guided LASIK (Active Comparator): Wavefront-guided LASIK
  Interventions: Procedure: Photorefractive keratectomy; Procedure: Laser in-situ keratomileusis

INTERVENTIONS:
Procedure: Photorefractive keratectomy — One eye undergoes wavefront-guided PRK with the Visx S4 CustomVue excimer laser.
  Other Names: PRK, CustomVue, Wavefront-guided
Procedure: Laser in-situ keratomileusis — One eye undergoes wavefront-guided LASIK using the Visx S4 excimer laser.
  Other Names: LASIK, CustomVue, Visx, Intralase FS60

SUMMARY:
A prospective comparison of eyes undergoing wavefront-guided LASIK in one eye and wavefront-guided PRK in their fellow eye for myopia.

DETAILED DESCRIPTION:
This is a research study comparing the outcomes of LASIK surgery to PRK surgery for nearsightedness when using the two different procedures. You will have one eye treated with LASIK using the Intralase FS laser and your other eye treated with PRK. You will be one of 100 sighted patients at Stanford to undergo treatment in this clinical research trial. This will be a prospective, randomized, research study in which up to 200 consecutive eyes scheduled to undergo excimer laser in situ keratomileusis (LASIK) in one eye and photorefractive keratectomy (PRK) in the fellow eye for the correction of myopia (nearsightedness) with or without astigmatism will be enrolled. The choice of which eye receives LASIK and which eye receives PRK will be randomized prior to enrollment. Randomization will be done according to a randomization schedule. You will know which eye is being treated with which procedure. The randomization will determine only whether your right or left eye is treated with the LASIK procedure. The other eye will be treated with PRK. You have a fifty percent chance of having your left eye treated with LASIK as your right eye. Subjects will undergo either bilateral (both eyes at once) wavefront (a more precise custom laser system) guided LASIK and PRK treatments using the VISX Star S4 excimer laser. All subjects will be followed for one year after the vision correction procedure. Subjects scheduled to undergo LASIK and PRK for the correction of myopia (nearsightedness) with or without astigmatism will be screened for eligibility. Eligible subjects will be examined preoperatively to establish a baseline for ocular condition (the general health and glasses prescription of the eyes). Postoperatively, subjects will undergo an ophthalmic evaluation (complete eye examination) at regular intervals as specified in this protocol. Retreatments (a second operation on the same eye for residual nearsightedness) will not be allowed during the first six months of this study. If you elect to undergo a retreatment of your LASIK or PRK surgery prior to the 6-month post-operative visit, the retreated eye will be exited from the study as of the retreatment date.

Any significant new finding developed during the course of the research which may relate to the subject's willingness to continue participation will be provided to the subject or subject's representative in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -0.75 diopters and -7.00 diopters with or without astigmatism of up to -3.50 diopters.

Exclusion Criteria:

* Subjects under the age of 21.
* Patients with thin corneas.
* Patients with topographic irregularities.
* Patients with keratoconus.
* Patients with autoimmune diseases.
* Patients who are pregnant or nursing.
* Patients must have similar levels of nearsightedness in each eye. They can not be more than 1.0 diopter of difference between eyes.
* Patients must have similar levels of astigmatism in each eye. They can not have more than 1.0 diopter of difference between eyes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Improvement in uncorrected visual acuity | Baseline to one year
Changes in best spectacle corrected visual acuity | Baseline to one year
Changes in 25 and 5% low contrast acuity | baseline to one year

SECONDARY OUTCOMES:
Changes in quality of vision | baseline to one year
Comparison of dry eye signs and symptoms between LASIK and PRK | baseline to one year
Changes in higher order aberrations | Baseline to one year

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Manche EE, Haw WW. Wavefront-guided laser in situ keratomileusis (Lasik) versus wavefront-guided photorefractive keratectomy (Prk): a prospective randomized eye-to-eye comparison (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2011 Dec;109:201-20. PMID 22253488